CLINICAL TRIAL: NCT02665533
Title: Evaluation of Two Pharmacological Protocols for Pre-emptive Analgesia in Impacted Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1.354.720
Record Dates: First submitted 2016-01-20; First posted 2016-01-27 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-01

CONDITIONS: Pain; Edema; Trismus
Keywords: pain measurement; edema; trismus
MeSH Terms: conditions — Pain; Edema; Trismus | interventions — Dexamethasone; dexamethasone acetate; Codeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Active Comparator): Dexamethasone 8 mg, one capsule single preoperative dose.
  Interventions: Drug: Dexamethasone
- Diclofenac Sodium associated with Codeine (Experimental): Diclofenac Sodium 50 mg associated with Codeine 50 mg, one capsule single preoperative dose.
  Interventions: Drug: Diclofenac Sodium associated with Codeine

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 8 mg
  Other Names: Dexamethasone Acetate
  Arms: Dexamethasone
Drug: Diclofenac Sodium associated with Codeine — Diclofenac Sodium 50 mg associated with Codeine 50 mg
  Arms: Diclofenac Sodium associated with Codeine

SUMMARY:
The main aim of the study is to investigate the pre-emptive effect of dexamethasone and diclofenac associated to codeine to prevent the pain, edema and limited mouth opening at the extraction of third molar.

DETAILED DESCRIPTION:
The surgery of third molar is usually associated with important post-surgical sequelae. The damage caused to tissue and bone may result in considerable pain, edema and trismus. The symptoms start gradually, peaking in 2 days after the extraction. The use of medications such as dexamethasone and diclofenac associated to codeine may support the prevention of post-surgical pain. This clinical trial aim compare the the pre-emptive effect of dexamethasone and diclofenac associated to codeine to prevent the pain, edema and limited mouth opening at the extraction of third molar.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication of asymptomatic bilateral extractions of lower third molars;
* Aged 18 years or older;
* Have a good health and no disease;

Exclusion Criteria:

* Patients with history of any medication treatment within 15 days before the beginning of the research, history of allergy to the drugs, substances or materials used in this study, pregnancy or lactation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Post-surgical swelling of third molar extraction determined using linear measures in the face | Up to seven days post-surgical
  During the post-surgical intervals of 24, 48 and 72 hours and seven days, the swelling was determined using linear measures in the face.
Post-surgical trismus of third molar extraction determined by maximum mouth opening | Up to seven days post-surgical
  During the post-surgical intervals of 24, 48 and 72 hours and seven days, the trismus was determined by maximum mouth opening.
Post-surgical pain of third molar extraction using visual analogic scale | Up to seven days post-surgical
  The post-surgical pain was self-recorded by the patient using visual analogic scale in intervals of 24, 48 and 72 hours and seven days.

SECONDARY OUTCOMES:
Analgesic consumption | Up to seven days post-surgical
Duration of surgery | Up to seven days post-surgical

CONTACTS AND LOCATIONS:
Overall Officials: Thiago Lima, Principal Investigator — Federal University of the Valleys of Jequitinhonha and Mucuri
Locations (1):
- Universidade Federal dos Vales do Jequitinhonha e Mucuri, Diamantina, Minas Gerais, Brazil